CLINICAL TRIAL: NCT02651038
Title: Pharmacokinetics of Micafungin During Continuous Venovenous Hemofiltration
Acronym: Mica-HDF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Florian Thalhammer, Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mica_HDF
Record Dates: First submitted 2015-07-17; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Candida Sepsis
MeSH Terms: interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Micafungin (Experimental): Micafungin is administered per clinical need and the pharmacokinetic parameters are analyzed
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — Measurement of PK

SUMMARY:
Micafungin is a cyclic lipopeptide antifungal agent of the echinocandin class. Members of this class of antifungal agents are known to inhibit the synthesis of glucan polymers in fungal cell walls. The spectrum of activity of micafungin includes Candida (all species, including strains resistant to fluconazole), Aspergillus, and Pneumocystis.

In intensive care patients continuous venovenous haemodiafiltration (CVVHDF) is a well-established extracorporal renal replacement therapy with a high clearance rate.

Pharmacokinetic studies of antifungal agents in critically ill patients treated with CVVHDF are rare. Elimination of any given drug by renal replacement therapy is determined by several major factors which are membrane specific, due to physico-chemical properties of the drug and characteristics of the renal replacement technique used.

Ten intensive-care patients with acute renal failure and suspected or proven candida infection are included into the study.

100 mg Micafungin will be infused over a period of sixty minutes via a central venous catheter, different from the venous catheter used for CVVHDF. Blood samples will be drawn on days 1 and 2 from the arterial and venous line of the extracorporeal circuit at 0, 2, 4, 6, 8 and 24h after starting the infusion. Plasma and ultrafiltration samples, collected from the outlet of the ultrafiltrate compartment of the hemofilter, will be taken at corresponding times.

The following pharmacokinetic parameters will be determined: area under the curve (AUC), half-live (t1/2), maximum plasma concentration (Cmax) and elimination fraction.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 70 years
* Suspected or proven candida infection requiring parenteral antifungal therapy.
* Continuous venovenous hemo(dia)filtration or Cica HD because of an acute renal failure.

Exclusion Criteria:

* Known history of hypersensitivity to echinocandins.
* An expected survival of less than three days.
* Known alcohol dependency
* Known epilepsy
* Known pregnancy
* Known liver failure
* Soor oesophagitis

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Haemofiltration clearance of Micafungin | 49 hours
  Haemofiltration clearance in ml/min measured by micafungin concentration gradient between hemodialyzer inlet and outlet port.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Thalhammer, Prof. Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Vossen MG, Knafl D, Haidinger M, Lemmerer R, Unger M, Pferschy S, Lamm W, Maier-Salamon A, Jager W, Thalhammer F. Micafungin Plasma Levels Are Not Affected by Continuous Renal Replacement Therapy: Experience in Critically Ill Patients. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e02425-16. doi: 10.1128/AAC.02425-16. Print 2017 Aug. PMID 28584142